CLINICAL TRIAL: NCT05921838
Title: The Role of Circ0014614 in the Formation and Development of ET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-173
Record Dates: First submitted 2023-05-31; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Primary Thrombocytosis
MeSH Terms: conditions — Thrombocythemia, Essential

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- ET patients: patients suffer from primary thrombocytosis
- healthy doner: Healthy individuals without blood system diseases

INTERVENTIONS:
Other:

SUMMARY:
Research on the Role of Circ0014614 in the Formation and Development of ET

DETAILED DESCRIPTION:
In recent years, tumor niche involved in the development of myeloproliferative disease（MPN）, which is remodelled by stem progenitor cells driving gene mutation, has attracted attention, but the reason and mechanism of remodelling microenvironment by mutated hematopoietic stem cells（ HSCs） are poorly understood. Our previous studies have shown that there is an obstacle in the transport of extracellular vesicles circ0014614 from MEPs in ET patients, which is enriched in the cytoplasm of megakaryocyte-erythroid progenitor（MEPs）, causing abnormal proliferation and reduced apoptosis of MEPs. The amplified MEPs affect the ossification of Mesenchymal stem cells（MCSs）. Based on this, we propose a hypothesis that circ0014614 may cause abnormal amplification of MEPs, reshape niche, induce ossification of MCSs, and abnormal amplification of osteoblasts（OBCs） through a certain pathway, promoting the formation and development of ET. This study will expand the collection of bone marrow samples from Essential thrombocytosis（ET） patients, detect the differences in circ0014614 levels in peripheral blood and bone marrow before and after treatment, and predict its downstream microRNA and mRNA through bioinformatics analysis to speculate its role in the occurrence and development of the disease. In recent years, tumor niche involved in the development of MPN, which is remodelled by stem progenitor cells driving gene mutation, has attracted attention, but the reason and mechanism of remodelling microenvironment by mutated HSCs are poorly understood. Our previous research has shown that there is an obstacle in the transport of extracellular vesicles circ0014614 from MEPs in ET patients, which is enriched in the cytoplasm of MEPs, causing abnormal proliferation and reduced apoptosis of MEPs. The amplified MEPs affect the ossification of MCSs. Based on this, we propose a hypothesis that circ0014614 may cause abnormal amplification of MEPs, reshape niche, induce ossification of MCSs, and abnormal amplification of OBCs through a certain pathway, promoting the formation and development of ET. This study will expand the collection of bone marrow samples from ET patients, detect the differences in circ0014614 levels in peripheral blood and bone marrow before and after treatment, and predict its downstream microRNA and mRNA through bioinformatics analysis to speculate its role in the occurrence and development of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. According to the classification and diagnostic criteria of hematological myeloid tumors by WHO 2016, patients diagnosed as ET are standardized
2. Voluntary signing of informed consent form
3. Age ≥ 18 years old, regardless of gender
4. No pregnancy plan during treatment

Exclusion Criteria:

1.The researcher judged that it was not suitable to participate in this study

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: ET patients treated with interferon
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Circ0014614 copies in ET patients treated with interferon for 8 months | 8months
  Circ0014614 copies in ET patients treated with interferon for 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Dan Xu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No